CLINICAL TRIAL: NCT02124525
Title: The Efficacy of N-acetylcysteine as a Cessation Treatment for Tobacco Smoking and Oxidative Stress Reduction
Brief Title: N-acetylcysteine for Tobacco Smoking
Acronym: NACNOS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Eduardo Salviano Teixeira Prado, MD, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UEL 33553/2011
Record Dates: First submitted 2013-01-13; First posted 2014-04-28 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Tobacco Smoking; Oxidative Stress; Inflammation
MeSH Terms: conditions — Tobacco Smoking; Inflammation | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-acetylcysteine (Placebo Comparator): Subjects receiving N-acetylcysteine (NAC): 6 pills/ day of N-acetylcysteine 500mg.
  Duration: 12 weeks
  Interventions: Drug: N-acetylcysteine
- Placebo (Placebo Comparator): Placebo will be taken for 12 weeks

INTERVENTIONS:
Drug: N-acetylcysteine — N-acetylcysteine 3000mg a day for 12 weeks versus Placebo for 12 weeks
  Other Names: N-acetylcysteine 3000mg a day for 12 weeks
  Arms: N-acetylcysteine

SUMMARY:
The purpose of this study is to investigate the efficacy of N-acetylcysteine (NAC) for smoking cessation in a double blind, randomized, placebo-controlled trial. Simultaneously, the study aims to elucidate the role of inflammatory markers and oxidative stress related to nicotine addiction and the use of NAC, an acetylated precursor of cysteine, a naturally occurring amino acid that has antioxidant actions in its own right, in reducing oxidative stress and inflammation in smokers. It will evaluate the use of NAC in smoking cessation, after 4, 8 and 12 weeks of treatment.

DETAILED DESCRIPTION:
The study will be conducted at the Center of Smoking Cessation, at State University (UEL), in Brazil. A sample of 32 outpatients will be selected, that are refractory to first-line smoking cessation treatment. All patients included in this study under the condition of understanding and signing the informed consent after approval of the research by Ethics Research Committee of UEL. Prior to randomization into the clinical trial, all participants will be assessed with a questionnaire to provide information about demographic, smoking history, nicotine dependence, depressive disorder, anthropometric measurements such as , height, weight, body mass index (BMI), waist circumference (WC), as well as heart rate (HR) and blood pressure (BP).The diagnostic criteria for research for depressive disorder and tobacco use disorder will be assed by trained psychiatrists according to the Structured Clinical Interview. The primary outcome measurement will be the significant reduction on the number of cigarettes/day. Secondary outcome measurements will be: reduction on the exhaled Carbon Monoxide, reduction of Hamilton Depression Rating Scale scores, improvement on Sheehan Quality of Life scale measurements.

The Fagerstrom Test for nicotine dependence (FTND) will be used to assess the severity of tobacco by dependence FTND. The FTND has a scale of six items and the score 0-10. The cutoff point for FTND nicotine dependence will be > 5. The assessment of severity of depression among study participants will be conducted by using Hamilton Depression Rating Scale- 17 items (HDRS). HDRS was translated and adapted for the Brazilian population. Minnesota Nicotine Withdrawal Scale (MNWS) MNWS is a 5-point scale (none, slight, mild, moderate, severe) to measure withdrawal symptoms.The scale assesses the damage that the patient is having due to illness. It is a self - administered scale consisting of 3 items. A score of 0-10 corresponds to the patient's opinion. Assesses the disability damage in three areas: 1) occupational, 2) social life, leisure, 3) family life, activities, and household activities. Can be scored 0-10, 0-3 mild injury, 4-6 moderate damage and 7-10 injury grave.The number of pack-years was calculated according to the definition: the number of cigarettes smoked per day multiplied by number of years smoked and divided by 20 (1 pack has 20 cigarettes).This clinical trial was designed to investigate the efficacy of NAC as a treatment for tobacco use disorder. Data were collected by face-to-face interview at baseline and weeks 4, 8 and 12. Smoking status was also evaluated using exhaled carbon monoxide (COEXH). COEXH was measured using a Micro CO Meter with an electrochemical sensor (Micro CO - Micro Medical Ltd, Rochester, Kent, UK). All participants were instructed to breathe deeply and to hold their breath for 20 seconds and then to exhale slowly and completely through a mouthpiece. Smoking reduction was validated by breath carbon monoxide concentration, and the cut-off point for COEXH levels will be categorized as ≤ 6ppm for smoking cessation (Middleton et al., 2000). Both groups will receive monthly meetings of Group Behavioral Therapy during the course of the study.

Participants (n=32) were randomized into two groups 16 patients in each group, in a double-blind manner to receive NAC or placebo. The dose of NAC was 3000mg/day administered in 500 mg capsules in two daily doses, 3 capsules in the morning and 3 in the evening. The chosen dosage was based on previous studies in which similar dosages had shown to be effective and well tolerated.

Individuals were randomized to NAC or placebo, each group have individuals with equal gender, age, scores of FTND and depressive disorders.

Statistical analysis will be performed with repeated measurements design analyses of variance, and post hoc t test.

ELIGIBILITY:
Inclusion Criteria:

* Current daily smoker of 10 or more cigarettes per day
* Capacity to consent to the study and follow its instructions and procedures
* Female participants will need to be utilizing effective contraception if of childbearing age
* Must be able to swallow the pills

Exclusion Criteria:

* Clinically unstable medical or psychiatric disorders that require acute treatment
* Active gastrointestinal ulcers
* Pregnancy or breastfeeding
* Current use of vitamin supplements or other substances with recognized antioxidant action
* A history of anaphylactic reaction to NAC or any component of the preparation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-04 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
The efficacy of N-acetylcysteine in reducing of the cigarettes per day | At Baseline and after 12 weeks (endpoint)
  The primary outcome will be the significant reduction of the cigarettes per day

SECONDARY OUTCOMES:
Efficacy of N-acetylcysteine in reducing exhaled Carbon Monoxide | At Baseline and after 12 weeks (endpoint)
  The secondary outcomes will be the significant reduction of the exhaled Carbon Monoxide

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Nunes, MD, PhD, Principal Investigator — Londrina State University - Center of Smoking Cessation
Locations (1):
- Hospital das Clínicas da Universidade Estadual de Londrina (Londrina State University Clinical Hospital), Londrina, Paraná, Brazil